CLINICAL TRIAL: NCT03095157
Title: The Emerging Role of Resolvins in the Prevention of Chronic Pain After Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Mieke A. Soens, MD Staff Anesthesiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017P000346
Record Dates: First submitted 2017-03-16; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Patients Scheduled for Thoracic Surgery/Esophagectomy Will be Enrolled; Persistent Post Surgical Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: fractionated marine lipid concentrate derived from anchovy and sardine oil
- Treatment (Experimental)
  Interventions: Dietary Supplement: fractionated marine lipid concentrate derived from anchovy and sardine oil

INTERVENTIONS:
Dietary Supplement: fractionated marine lipid concentrate derived from anchovy and sardine oil — Patients will be randomized to receive perioperative treatment versus placebo

SUMMARY:
The aim of the study is to investigate whether pre-operative dysregulated systemic lipid mediator pathways are associated with increased risk for the development of persistent post surgical pain. In addition we will investigate whether treatment with an over the counter dietary supplement containing a fractionated marine lipid derivative from anchovy and sardine oil prevents the development of chronic pain after surgery.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo esophagectomy at BWH
* 18-80 years old

Exclusion Criteria:

* pre-existing chronic pain
* current opioid use
* current treatment with corticosteroids
* evidence of active infection
* chronic liver disease
* end-stage renal disease (CKD-5)
* chronic inflammatory disorders
* recent major surgery or illness within 30 days
* use of immunosuppressive medication
* history of organ transplant
* pregnancy or plans to become pregnant
* lactating
* allergies to fish or fish oil

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Primary Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (0=no pain; 10=worst imaginable pain) at 3 months after surgery | 3 months
  Persistent pain after thoracic surgery

IPD SHARING:
Plan to Share IPD: No